CLINICAL TRIAL: NCT01513967
Title: A Randomized Single and Multiple Dose Study Evaluating the Safety and Tolerability of RPh201 in Healthy Subjects and in Adults With Alzheimer's Disease
Brief Title: A Randomized SAD and MAD Study Evaluating the Safety and Tolerability of RPh201 in Healthy Subjects and in Adults With Alzheimer's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regenera Pharma Ltd (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RGN-ADC-001
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Healthy Volunteers; Moderate to Severe Alzheimer Patients
Keywords: Alzheimer,; dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Part A, SAD Treatment 1 (Experimental): RPh201 single dose (SAD Low Dose )
  Interventions: Drug: RPh201, botanical drug product
- Part A, SAD Placebo 1 (Placebo Comparator): Placebo single dose (SAD Low Dose )
  Interventions: Drug: Placebo
- Part A, SAD Treatment 2 (Experimental): RPh201 single dose (SAD Mid Dose )
  Interventions: Drug: RPh201, botanical drug product
- Part A, SAD Placebo 2 (Placebo Comparator): Placebo single dose (SAD Mid Dose )
  Interventions: Drug: Placebo
- Part A, SAD Treatment 3 (Experimental): RPh201 single dose (SAD High Dose )
  Interventions: Drug: RPh201, botanical drug product
- Part A, SAD Placebo 3 (Placebo Comparator): Placebo single dose (SAD High Dose )
  Interventions: Drug: Placebo
- Part B, MAD Treatment 1 (Experimental): RPh201 multiple dose (MAD Low Dose )
  Interventions: Drug: RPh201, botanical drug product
- Part B, MAD Placebo 1 (Placebo Comparator): Placebo multiple dose (MAD Low Dose )
  Interventions: Drug: Placebo
- Part B, MAD Treatment 2 (Experimental): RPh201 multiple dose (MAD Mid Dose )
  Interventions: Drug: RPh201, botanical drug product
- Part B, MAD Placebo 2 (Placebo Comparator): Placebo multiple dose (MAD Mid Dose )
  Interventions: Drug: Placebo
- Part B, MAD Treatment 3 (Experimental): RPh201 multiple dose (MAD High Dose )
  Interventions: Drug: RPh201, botanical drug product
- Part B, MAD Placebo 3 (Placebo Comparator): Placebo multiple dose (MAD High Dose )
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RPh201, botanical drug product — SC administration at varying doses
  Arms: Part A, SAD Treatment 1; Part A, SAD Treatment 2; Part A, SAD Treatment 3; Part B, MAD Treatment 1; Part B, MAD Treatment 2; Part B, MAD Treatment 3
Drug: Placebo — SC administration at varying doses
  Arms: Part A, SAD Placebo 1; Part A, SAD Placebo 2; Part A, SAD Placebo 3; Part B, MAD Placebo 1; Part B, MAD Placebo 2; Part B, MAD Placebo 3

SUMMARY:
This is a dual-centre, Phase I/IIa study, in healthy subjects and subjects with AD to investigate the safety, tolerability, cognitive, and behavioural effects of RPh201. The study will be divided into three parts: A, B, and C (NOT Performed)

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of RPh201 after single and multiple ascending doses. This study is designed with sufficient time in between dose escalations to allow for an interim analysis of safety and tolerability data as this is considered the safest approach to assess the effects of a compound with an undefined mechanism and therapeutic target.

This protocol is written with some flexibility to accommodate the inherent dynamic nature of Phase I clinical studies. Modifications to the dose, dosing regimen, and/or clinical or laboratory procedures currently outlined below may be required to achieve the scientific goals of the study objectives and/or to ensure appropriate safety monitoring of the study subjects. Interim safety analyses will guide dose escalation/reduction in the trial.

ELIGIBILITY:
For PART A AND PART B (healthy volunteers, SAD and MAD)

Inclusion Criteria:

* healthy male or female subjects 18 to 65 years of age, inclusive
* body mass index (BMI) within the range of 18.0 to 33.0 kg/m2, inclusive, and a minimum weight of at least 50.0 kg at Screening
* female subjects of childbearing potential must be practicing abstinence or using and willing to continue using two medically acceptable form of birth control for at least 1 month prior to Screening (at least 3 months for oral and transdermal contraceptives) and for at least 1 month after the last study drug administration. Medically acceptable forms of contraception include oral or patch hormonal contraceptives, intrauterine device, progestin implant or injection, bilateral tubal ligation, or double-barrier (i.e., male condom in addition to a diaphragm or a contraceptive sponge).
* female subjects of non-childbearing potential must be amenorrheic for at least 2 years or had a hysterectomy and/or bilateral oophorectomy/salpingo-oophorectomy (as determined by subject medical history)
* male subjects of reproductive potential with a partner(s) of childbearing potential, must be using and willing to continue to using two medically acceptable contraceptive precautions from Screening and for at least 1 month after the last study drug administration. Medically acceptable forms of contraception include abstinence, vasectomy, or male condom for subjects
* female subjects must have a negative pregnancy test
* able to speak, read, and understand English sufficiently to understand the nature of the study, to provide written informed consent, and to allow completion of all study assessments
* must understand and provide written informed consent prior to the initiation of any protocol-specific procedures
* must be willing and able to abide by all study requirements and restrictions

Exclusion Criteria:

* current drug or alcohol dependence (excluding caffeine), based on self-report, including subjects who have been in a drug rehabilitation program
* current smoker or a history of using tobacco products within 3 months prior to Screening
* clinically significant abnormalities on physical examination, medical history, 12-lead ECG (i.e., QTc > 440 for male subjects and > 450 for female subjects), vital signs, or laboratory values, as judged by the investigator or designee
* history or presence of any clinically significant illness (e.g., cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, musculoskeletal, or psychiatric) or any other condition, which in the opinion of the investigator would jeopardize the safety of the subject or the validity of the study results
* use of a non-prescription drug within 7 days prior to the first drug administration. Subjects who have taken over-the-counter medication may still be entered into the study, if in the opinion of the investigator or designee, the medication received will not interfere with the study procedures or data integrity or compromise the safety of the subject
* use of any prescription medications, recreational drugs, or natural health products (except vitamin or mineral supplements, acceptable forms of birth control, and hormone replacement) within 14 days prior to first drug administration or throughout the study, unless in the opinion of the investigator or designee, the product will not interfere with the study procedures or data integrity or compromise the safety of the subject
* positive urine drug screen
* positive breath alcohol test. If a subject presents with positive breath alcohol test, the subject may be rescheduled at the discretion of the investigator or designee
* female subjects who are currently pregnant or lactating or who are planning to become pregnant within 60 days of last study drug administration
* history of allergy or hypersensitivity to mastic or related drugs (e.g., mastic gum, mastic resin, Chios mastic powder, retsina wine, Mastic Gum 500, Mastic Gum Elma 50, Nutricology Mastic Gum)
* history of allergy or hypersensitivity to cottonseed oil
* positive for Hepatitis B, Hepatitis C, or HIV
* current or pending legal charges or currently on probation
* treatment with any investigational drug within 30 days prior to first drug administration in the treatment phase
* a subject who, in the opinion of the investigator or designee, is not considered to be suitable and is unlikely to comply with the study protocol for any reason

For PART C (subjects with Alzheimer's Disease)

Inclusion Criteria:

* males and females ages ≥ 55 years of age at Screening visit
* diagnosis of AD, consistent with criteria from both the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) Criteria for Probable AD and Diagnostic and Statistical Manual of Mental Disorders - IV TR (DSM-IV TR) Criteria for Dementia of the Alzheimer's Type
* Mini-Mental Status Evaluation (MMSE) score of 5-15, inclusive, at Screening visit
* Rosen-Modified Hachninski Ischemia score of ≤ 4 at Screening visit
* subjects and caregivers must be able to read, write, and speak the language in which psychometric tests are provided with acceptable visual and auditory acuity
* subject must have a reliable informant (caregiver) to provide collateral history and who will facilitate the subject's full participation in the study
* subject and caregivers must provide written informed consent and be willing to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures
* subjects may continue on background cholinesterase inhibitor and/or memantine
* subjects must be in satisfactory good health, in the opinion of the investigator, based on medical history, physical examination, vital signs, 12-lead ECG, and laboratory tests
* magnetic resonance imaging (MRI) or computed tomography (CT) within 12 months of Screening visit consistent with a diagnosis of Probable AD without any other clinically significant findings

Exclusion Criteria:

* diagnosis or history of other dementia or neurodegenerative disorders causing cognitive impairment (e.g., Parkinson's disease, Lewy body disease, Fronto-temporal Dementia, alcohol and drug abuse, Traumatic Brain Injury).
* subjects receiving immunosuppressants, tricyclic anti-depressants, anticoagulants, or chemotherapeutic agents
* hypertension not adequately controlled, per investigator's judgment
* poorly controlled Type 1 and/or Type 2 diabetes, per investigator's judgment
* women of child bearing potential who are not using an effective method of birth control
* any other medical condition or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or that may interfere with the interpretation of study results, and that, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Faulknor, MD, Principal Investigator — Kendle Early Stage - Toronto; Sharon Cohen, MD, Principal Investigator — Toronto Memory Program
Locations (2):
- Canada (2):
  - Toronto Memory Program, Toronto, Ontario
  - Kendle Early Stage - Toronto, Toronto, Ontario

REFERENCES:
- [Result] Hazan Z, Adamsky K, Lucassen A, Levin LA. A First-in-Human Phase 1 Randomized Single and Multiple Ascending Dose Study of RPh201 in Healthy Volunteers. Clin Pharmacol Drug Dev. 2020 Apr;9(3):366-374. doi: 10.1002/cpdd.720. Epub 2019 Jun 28. PMID 31250992

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A, SAD Treatment 1 5mg: RPh201 single dose (SAD 5mg)
  RPh201, botanical drug product: SC administration at varying doses
- Part A, SAD Treatment 2: RPh201 single dose (SAD 10mg)
  RPh201, botanical drug product: SC administration at varying doses
- Part A, SAD Treatment 3: RPh201 single dose (SAD 20mg)
  RPh201, botanical drug product: SC administration at varying doses
- Part A, SAD Placebo: Placebo single dose (SAD 20mg)
  Placebo: SC administration at varying doses
- Part B, MAD Treatment 1: RPh201 multiple dose (MAD 5mg)
  RPh201, botanical drug product: SC administration at varying doses
- Part B, MAD Treatment 2: RPh201 multiple dose (MAD 10mg)
  RPh201, botanical drug product: SC administration at varying doses
- Part B, MAD Treatment 3: RPh201 multiple dose (MAD 20mg)
  RPh201, botanical drug product: SC administration at varying doses
- Part B, MAD Placebo: Placebo multiple dose (MAD 20mg)
  Placebo: SC administration at varying doses
Period: Overall Study
Arm/Group | Part A, SAD Treatment 1 5mg | Part A, SAD Treatment 2 | Part A, SAD Treatment 3 | Part A, SAD Placebo | Part B, MAD Treatment 1 | Part B, MAD Treatment 2 | Part B, MAD Treatment 3 | Part B, MAD Placebo
Started | 4 | 4 | 4 | 6 | 4 | 4 | 5 | 8
Completed | 4 | 4 | 4 | 6 | 4 | 3 | 3 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — missed a study visit | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — excluded due to positive drug screen | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part C of the study has not been initiated
Groups:
- Part A, SAD Treatment 1 (5mg): RPh201 single dose (SAD 5mg)
  RPh201, botanical drug product: SC administration at varying doses
- Part A, SAD Treatment 2 (10mg): RPh201 single dose (SAD 10mg)
  RPh201, botanical drug product: SC administration at varying doses
- Part A, SAD Treatment 3 (20mg): RPh201 single dose (SAD 20mg)
  RPh201, botanical drug product: SC administration at varying doses
- Part A, SAD Placebo: Placebo single dose (SAD)
  Placebo: SC administration at varying doses
- Part B, MAD Treatment 1 (5mg): RPh201 multiple dose (MAD 5mg)
  RPh201, botanical drug product: SC administration at varying doses
- Part B, MAD Treatment 2 (10mg): RPh201 multiple dose (MAD 10mg)
  RPh201, botanical drug product: SC administration at varying doses
- Part B, MAD Treatment 3 (20mg): RPh201 multiple dose (MAD 20mg)
  RPh201, botanical drug product: SC administration at varying doses
- Part B, MAD Placebo: Placebo multiple dose (MAD)
  Placebo: SC administration at varying doses
- Total: Total of all reporting groups
Arm/Group | Part A, SAD Treatment 1 (5mg) | Part A, SAD Treatment 2 (10mg) | Part A, SAD Treatment 3 (20mg) | Part A, SAD Placebo | Part B, MAD Treatment 1 (5mg) | Part B, MAD Treatment 2 (10mg) | Part B, MAD Treatment 3 (20mg) | Part B, MAD Placebo | Total
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 4 | 4 | 5 | 8 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 6 | 4 | 4 | 5 | 8 | 39
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 39.8 [27 to 52] | 48.8 [38 to 65] | 50.8 [38 to 58] | 43.0 [32 to 54] | 42.5 [34 to 58] | 43.0 [23 to 60] | 40.8 [30 to 51] | 44.1 [22 to 63] | 44.0 [22 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 2 | 2 | 3 | 2 | 6 | 19
  Male | 1 | 3 | 4 | 4 | 2 | 1 | 3 | 2 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 3 | 1 | 0 | 1 | 2 | 11
  Not Hispanic or Latino | 3 | 3 | 2 | 3 | 3 | 4 | 4 | 6 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 7
  White | 2 | 4 | 3 | 5 | 4 | 2 | 4 | 5 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 4 | 4 | 6 | 4 | 4 | 5 | 8 | 39
BMI (kg/m2) [Mean (Full Range); unit: (kg/m2)] | 24.03 [22.1 to 26.7] | 26.01 [23.9 to 30.5] | 28.75 [26.1 to 32.1] | 25.04 [22.6 to 27.3] | 26.83 [23.4 to 28.6] | 23.60 [21.7 to 26.7] | 26.72 [23.3 to 29.2] | 25.36 [21.0 to 28.4] | 25.7 [21.0 to 32.1]
Height [Mean (Full Range); unit: cm] | 168.0 [163 to 175] | 169.5 [162 to 185] | 169.9 [159 to 178] | 168.2 [161 to 177] | 168.2 [160 to 175] | 162.5 [157 to 165] | 166.9 [160 to 181] | 164.3 [158 to 180] | 166.9 [157 to 185]
Weight [Mean (Full Range); unit: kg] | 67.7 [64 to 74] | 75.7 [66 to 104] | 82.8 [76 to 91] | 70.8 [66 to 83] | 75.8 [70 to 87] | 62.2 [59 to 66] | 74.3 [62 to 83] | 68.5 [52 to 75] | 71.8 [52 to 104]

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective: to Evaluate the Safety and Tolerability of RPh201 After Single and Multiple Rising Doses.
Description: Safety and tolerability following single and multiple ascending SC injection doses as assessed by Treatment-Emergent Adverse Events
Time Frame: up to 1 month
Population: The study analysis populations included the following:
  Randomized Population: All subjects who were assigned a randomization number in the Treatment Phase.
  Safety Population: All randomized subjects who received any study treatment in the Treatment Phase.
Measure: Count of Participants; unit: Participants
Groups:
- Part A, SAD Treatment 5mg: RPh201 single dose (SAD Low Dose )
  RPh201, botanical drug product: SC administration at varying doses
- Part A, SAD Treatment 10mg: RPh201 single dose (SAD Mid Dose )
  RPh201, botanical drug product: SC administration at varying doses
- Part A, SAD Treatment 20mg: RPh201 single dose (SAD High Dose )
  RPh201, botanical drug product: SC administration at varying doses
- Part A, SAD Placebo: Placebo single dose (SAD High Dose )
  Placebo: SC administration at varying doses
- Part B, MAD Treatment 5mg: RPh201 multiple dose (MAD Low Dose )
  RPh201, botanical drug product: SC administration at varying doses
- Part B, MAD Treatment 10mg: RPh201 multiple dose (MAD Mid Dose )
  RPh201, botanical drug product: SC administration at varying doses
- Part B, MAD Treatment 20mg: RPh201 multiple dose (MAD High Dose )
  RPh201, botanical drug product: SC administration at varying doses
- Part B, MAD Placebo: Placebo multiple dose (MAD High Dose )
  Placebo: SC administration at varying doses
Arm/Group | Part A, SAD Treatment 5mg | Part A, SAD Treatment 10mg | Part A, SAD Treatment 20mg | Part A, SAD Placebo | Part B, MAD Treatment 5mg | Part B, MAD Treatment 10mg | Part B, MAD Treatment 20mg | Part B, MAD Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 4 | 4 | 5 | 8
Participants
  Subjects with TEAE | 2 | 2 | 1 | 2 | 3 | 4 | 4 | 4
  Subjects with SAE | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Subjects with study drug discontinued due to AE | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Part A - SAE. 24-hour post-dose. A Follow-up visit within 5 to 7 days, approximately, of the drug administration. Part B - MAD. 4 Weeks Treatment Phase. A Follow-up visit within 5 to 7 days, approximately, of their last drug administration.
Description: All AEs reported from the time of informed consent for study participation were recorded. The investigator or designee and research site staff were responsible for the detection, documentation, and reporting of events meeting the definition of an AE or SAE.
Arm/Group | Part A, SAD Treatment 1 (5mg) | Part A, SAD Treatment 2 (10mg) | Part A, SAD Treatment 3 (20mg) | Part A, SAD Placebo | Part B, MAD Treatment 1 (5mg) | Part B, MAD Treatment 2 (10mg) | Part B, MAD Treatment 3 (20mg) | Part B, MAD Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/6 | 0/4 | 0/4 | 1/5 | 0/8
Other Adverse Events (participants affected / at risk) | 2/4 | 2/4 | 1/4 | 2/6 | 3/4 | 4/4 | 4/5 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, SAD Treatment 1 (5mg) (N=4) | Part A, SAD Treatment 2 (10mg) (N=4) | Part A, SAD Treatment 3 (20mg) (N=4) | Part A, SAD Placebo (N=6) | Part B, MAD Treatment 1 (5mg) (N=4) | Part B, MAD Treatment 2 (10mg) (N=4) | Part B, MAD Treatment 3 (20mg) (N=5) | Part B, MAD Placebo (N=8)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, SAD Treatment 1 (5mg) (N=4) | Part A, SAD Treatment 2 (10mg) (N=4) | Part A, SAD Treatment 3 (20mg) (N=4) | Part A, SAD Placebo (N=6) | Part B, MAD Treatment 1 (5mg) (N=4) | Part B, MAD Treatment 2 (10mg) (N=4) | Part B, MAD Treatment 3 (20mg) (N=5) | Part B, MAD Placebo (N=8)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia oral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (11) | 1 (3) | 2 (3)
Injection site pain (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 4 (4) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 1 (7) | 1 (1) | 0 (0) | 0 (0)
Hypermetropia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Oral mucosal erthema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site anaethesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 2 (2) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less